CLINICAL TRIAL: NCT05682534
Title: Examination of Musculoskeletal System Problems and Affecting Factors in CrossFit Sports
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Merve Paksoy, physiotherapist, Eastern Mediterranean University
Other Study IDs: ETK00-2022-0231
Record Dates: First submitted 2022-12-25; First posted 2023-01-12 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: CrossFit
Keywords: Musculoskeletal; CrossFit; Injury; Relationship; Risk Factors
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the relationship between musculoskeletal system problems and physical risk factors in CrossFit athletes. Athletes who do CrossFit training in the Turkish Republic of Northern Cyprus and meet the inclusion criteria will be included in the study. Individuals will first be asked about their personal information, when they started CrossFit, and their previous injury information. Then, the muscle strength, functionality, stability, balance of the lower extremity muscles and body posture in different positions will be evaluated with the determined tests. Evaluations are in a single day and in total 45 minutes. is planned in.

DETAILED DESCRIPTION:
CrossFit was developed by Greg Glassman in 1995 to increase core strength and general muscle strength and conditioning. It has grown in popularity around the world since it was first developed. Today, more than 15,000 CrossFit gyms operate around the world. CrossFit; It is a multimodal exercise training performed at high intensity, covering many functional movement models in a single exercise session. CrossFit is done with high-intensity, functional movements called "Workout of the Day" (GA). In workouts, exercises are performed quickly, with little or no rest between reps and sets. CrossFit training, which focuses on constantly changing functional movements; olympic weightlifting, powerlifting, sprint, plyometric, calisthenics, gymnastics and rope climbing is a mix of exercise models that are difficult to categorize. Each GA has its own special name and is performed with a certain combination of exercises. Although the nature of each session varies between affiliates, each session is typically 1 hour and includes a specific work of warm-up, strength or skill technique. Although GAs are performed in groups, the warm-up or cool-down times may differ according to the needs of the individuals.

Ángel Rodríguez et al. In their study on the epidemiology of injury and risk factors in CrossFit in 2020, they reported that the risk of injury in these sports modalities is similar when compared to other weightlifting and powerlifting, but challenging training programs increase the risk, especially if not performed in the right position. They emphasized that excess exercise volume and number of training sessions in CrossFit can cause early fatigue, higher effort perception, and a risky movement practice.

Mehrab et al. In another study conducted in 2017, they examined the injury incidence of Dutch CrossFit athletes and the injury incidence of athletes participating in CrossFit was 56.1% and the most injured body parts were 28.7% shoulder, 15.8% waist and 8.3% knee. have reported. The most common exercises causing injury were squat 22.0% and deadlift 18.0%. It has been stated that advanced athletes are more seriously injured than beginner athletes, and people with 3 years of CrossFit experience are 3.3 times more likely to be injured than those with 2 years or less experience. According to the review of 2020, it is reported that tendinopathies, joint injuries and muscle injuries are seen most frequently in Crossfit.

Given the growing popularity of CrossFit, avoiding potential risks from poor practice and proper training are essential for athletes. Analysis of injury patterns is an essential part of this process, enabling athletes, coaches, and health professionals to become better informed about inappropriate habits that harm physical integrity and how it can be improved. When we look at the literature, there are few studies that determine the physical risk factors of CrossFit athletes, and there is no study that examines the relationship between musculoskeletal injuries and risk factors. Our study will be the first study to determine the relationship between musculoskeletal system problems and physical risk factors of CrossFit athletes in the TRNC. The risk factors that emerged as a result of the study will be shared with the athletes, and the prevention of possible future injuries and the improvement of public health will be tried.

Hypotheses:

H01: Balance is similar in CrossFit athletes with and without musculoskeletal system problems.

H02: Functional performance is similar in CrossFit athletes with and without musculoskeletal system problems.

H03: Stability is similar in CrossFit athletes with and without musculoskeletal system problems.

H04: Muscle strength is similar in CrossFit athletes with and without musculoskeletal system problems.

H05: Posture is similar in CrossFit athletes with and without musculoskeletal system problems.

Material and Method:

Athletes who do CrossFit training in the Turkish Republic of Northern Cyprus and meet the inclusion criteria will be included in the study. The sociodemographic information of the individuals and in addition to this information, the training characteristics of the individuals (daily training time, etc.), the time to start CrossFit will be questioned. Then, lower extremity muscle strength, function, posture in lateral and squat positions, upper and lower extremity stability and balance will be evaluated. Evaluations will be made within a single day.

In this study conducted to determine the relationship between musculoskeletal system problems and physical risk factors in CrossFit athletes; According to the power analysis using the G*Power program, in 2020 Lima et al. With reference to his study titled "Epidemiology and associated factors for CrossFit-related musculoskeletal injuries: a cross-sectional study", O.R. Its value was determined to be 2.25. Accordingly, the sample size required for 80% (1-β=0.95) power at α=0.05 level was calculated as 67 people. While 67 people participated in the evaluation, our study was completed with 65 people because 2 people who experienced health problems during the study left the study.

Evaluations to be applied to the Subject:

Socio-demographic Evaluations:

In the first evaluation, socio-demographic information such as age, height and body weight of individuals will be obtained through a form. In addition to this information, the training characteristics of the individuals (daily training time, etc.), the time to start CrossFit, the age of sports (how many years he has been training regularly) will be questioned.

Extended Nordic Musculoskeletal Questionnaire:

Turkish translation and cross-cultural adaptation Alaca et al. The Extended Nordic Musculoskeletal Questionnaire (GNSSA) is an assessment questionnaire used for the evaluation of musculoskeletal disorders. GNKİSA is a questionnaire that evaluates the presence, onset, incidence, results and effects of musculoskeletal pain in 9 regions of the body, including neck, shoulder, back, elbow, hand/wrist, waist, hip/thigh, knee, foot/ankle. . In this questionnaire, the age of onset of pain, hospitalization due to pain, changing the place of duty, having pain in the last year, last month and today are questioned. In addition, it is a questionnaire that can be filled by oneself or by interviewing the person, questioning whether the current pain affects the individual's work/home life, applying to a doctor/physiotherapist, taking medication and getting a report. Subjects are asked to mark the location of the pain on the body diagram. A high score indicates musculoskeletal pain.

Lower Extremity Functional Performance Evaluation:

Individuals' lower extremity functional performance will be evaluated with the Single Leg Jump Test (TBS). It is used in athletes and healthy young individuals in terms of being easy to use and not requiring equipment for the evaluation of functional performance during the return to sports phase. TBST validity and reliability were reported as 0.85 with ICC ratio. For the test, 2 measuring tapes are affixed to the plastic rods at an angle of 180 degrees and it is requested to stand on the dominant foot with the tip of the toe to the starting point of the tape measure. While the individual is standing on the dominant right leg, the other leg is bent at the knee and asked to jump forward and the point where the individual falls (heel projection) is marked. Care should be taken to keep the hands on the waist while jumping. If he loses his balance while falling to the ground and gets support from the other foot, the test is considered invalid and repeated. Jumping was repeated 3 times for both extremities. Jump distance is calculated by measuring with a tape measure in centimeters and taking the average value.

Evaluation of Lower Extremity Isokinetic Muscle Strength:

Strength values of isokinetic lower extremity quadriceps femoris and hamstring muscles will be measured by using an isokinetic dynamometer device (Humac Norm Isocynetic Dynanometer). In addition, the knee Q/H ratio will be calculated. Before starting the test, the test protocol will be explained in detail to the athletes and they will be warmed up with a 10-minute jog run. The movements of the athletes will be evaluated with a test protocol with 5 repetitions at 60º/sec and 20 repetitions at 180º/sec. A 1 minute rest will be given between measurements. Before each angular velocity, individuals are allowed to make 3 repetitive trials, and the tests will be applied after a rest period of 10 seconds. The test will be performed in a sitting position, the body will be positioned upright, the hips will be in 90° flexion, and the body and waist will be fixed in order to prevent compensation. Measurements to be applied in sitting position will be adjusted at 90° knee flexion and knee extension range of motion. The test will be applied bilaterally. total work; Joules (J) and peak torque will be recorded in Newtonmeters/kilogram (Nm/kg). In addition, the Shoulder Q/H ratio will be calculated.

Closed Kinetic Chain Upper Extremity Stability Test:

The reliability of the Closed Kinetic Chain Upper Extremity Stability Test was determined by Oliveira et al. made by Dynamic stability of the shoulder will be evaluated with KKZÜEST. This test, which is normally done in the push-up position, can be modified and applied in such a way that the knees are flexed for the elderly. The tester first explains the test position to the athlete, then the test is started with the 'start' command and the test is finished with the 'stop' command. After the instructions and demonstration, 3 trials are made to teach the test and 5 seconds rest between each trial. Verbal cues can be given as needed during practice. Subjects will be placed in a push-up position with their hands 36 inches (91.44 centimeters) apart on 1.5 inches (3.81 centimeters) wide strips. While one hand is fixed on the ground, it is asked to raise the other hand, touch the band under the fixed hand and take it back to the starting point. The same movement is repeated for the opposite side and 15 seconds. The number of repetitions performed is recorded. The test is performed 3 times and between trials, the participant is given 45 seconds. rest period is given. The average of 3 repetitions of the test is calculated using two formulas: test score and strength. The score is calculated as the average of 3 repetitions / height (m), Strength = 68% body weight (kg) x the average of 3 repetitions.

Closed Kinetic Chain Lower Extremity Stability Test:

Closed Kinetic Chain Lower Extremity Stability Test, Arıkan et al. Its reliability and validity were made in 2021 by The test was developed to measure trunk and lower extremity strength, strength and stability of the whole body. In addition, this test provides assessment of functional lower extremity stability, static/dynamic control of the lower extremity (knee/hip) or trunk, and simultaneous activation/such coactivation of the quadriceps and hamstring muscles. The tester first explains the test position to the athlete, then the test is started with the 'start' command and the test is finished with the 'stop' command. In order to teach the test from the instructions and demonstration, 3 trials are made and 5 seconds rest between each trial. Verbal cues can be given as needed during practice. A stable base floor, mat and stopwatch will be used as equipment to measure the test. (KKZAEST) starting position is on the mat on the stable floor, the person lies on his forearms with his feet shoulder-width apart, toes in contact with the floor and his body lies in a straight line. While maintaining the starting position of the body, the individual is asked to bring one foot to the diagonal outer side of the other foot. After touching the side of the other foot, the foot returns to the starting position. Then the person performs the same movement with the other foot. The number of repetitions in 15 seconds is recorded as in the closed kinetic chain upper extremity stability test. Touches count each time the foot touches the side of the other foot and the floor. Three repetitions of the 15-second CCZAEST are performed with 1-minute intervals between each test. The test is performed 3 times and between trials, the participant is given 45 seconds. rest period is given. The average of 3 repetitions of the test is calculated using two formulas: test score and strength. Score = average of 3 repetitions / average over height (m), Power = 68% body weight (kg) x average of 3 repetitions.

Upper Extremity Y Balance Test:

UEYDT is used to determine the risk of injury in musculoskeletal problems and is the only test in the literature that evaluates both shoulder stabilization and core stability. The tester first explains the test position to the athlete, and then 3 attempts are made to teach the test and rest for 5 seconds between each attempt. Verbal cues can be given as needed during practice. With both hands shoulder-width apart, the measurement begins with the right hand on the stance plate and the left hand on the access cursor. By maintaining the push-up position, the distance reached with the left hand is recorded in 3 directions, first medial, then inferolateral and finally superolateral. The person returns to the starting point in a controlled manner without breaking the push-up position. Tests are repeated 3 times on both extremities. Upper extremity length to be used in scoring is determined by measuring the distance between the acromion and the longest fingertip with a tape measure. The combined reach distance is calculated with the formula [(maximum medial + maximal inferolateral + maximal superolateral) / (3 x upper extremity length)] x 100 using the best value reached for both extremities in that direction.

Lower Extremity Y Balance Test:

Lower extremity dynamic balance will be evaluated with the Y Balance Test. Y balance test is a modified form of star balance test. The reliability of the test has been proven with ICC values varying between 0.85-0.91. The tester first explains the test position to the athlete, and then 3 attempts are made to teach the test and rest for 5 seconds between each attempt. Verbal cues can be given as needed during practice. In the test setup, 3 measuring tapes are adhered to the plastic rods at an angle of 120 degrees. Individuals stand on one leg at the intersection of the three measuring tapes. With the other foot, it is requested to extend the tip of the toe towards these 3 directions, anterior, posteromedial and posterolateral. At this time, care is taken to ensure that the individual does not lose his balance by placing his hands on his waist, that the heel of the foot he is standing on does not rise from the ground, and that the toes of the extended foot lightly touch the tape measure. At the end of each test, the individual is asked to bring his or her feet to the side without losing balance and without touching the ground. Measurements are repeated if the individual is unable to maintain one foot balance on the platform, or if the outstretched foot kicks the pointer plate or cannot return to the starting position. The test will be repeated 3 times in each direction and the average will be recorded in cm. The length of the lower extremity (between the spina iliaca anterior superior and the medial 3malleolus) will be measured with a tape measure. The combined reach distance will be calculated with the formula [(maximum anterior + maximal posteromedial + maximal posterolateral) / (3 x lower extremity length)] x 100 using the best value reached for both extremities in that direction.

Posture Evaluation:

Posture of the athletes in lateral and squat positions was reported by Hopkins et al. It will be measured with the PostureScreen Mobile® Application, whose validity and reliability study has been carried out by PostureScreen Mobile® Application is a valid and reliable application that allows individuals to evaluate their postures through photographs with the help of the camera system on devices with iOS and Android systems. The application, which provides the opportunity to evaluate the static posture of individuals in standing posture from the anterior, posterior and lateral aspects and the posture in the squat position from the lateral aspect, reports numerical deviations from normal posture. Postures of the athletes in lateral and squat positions will be done on the smartphone using the PostureScreen Mobile® App. The specific points determined in the application for the lateral and squat positions of the athletes will be marked using the touch screen on the photographs taken, and according to these points, the postural disorder values and the degree of the disorder will be calculated and reported for each variable in cm or degrees via the software.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 20-45
* Those who have been doing CrossFit sports for at least 1 year
* Those who do CrossFit at least 2 days a week

Exclusion Criteria:

* Those who train independently outside of CrossFit
* Those with neurological problems diagnosed by a doctor
* Those who received physiotherapy in the last 6 months

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Athletes in the Turkish Republic of Northern Cyprus who have done CrossFit sport for at least one year, who train at least 2 days a week and between the ages of 20-45 will be included in the study.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Isokinetic Muscle Strength Assessment | 5 months
  Quadriceps and hamstring muscle strengths will be evaluated with a test protocol with 5 repetitions at 60º/sec speed and 20 repetitions at 180º/sec speed.

SECONDARY OUTCOMES:
Extended Nordic Musculoskeletal Questionnaire | 5 months
  Turkish translation and cross-cultural adaptation Alaca et al. The Extended Nordic Musculoskeletal Questionnaire is an assessment questionnaire used for the evaluation of musculoskeletal disorders. İs a questionnaire that evaluates the presence, onset, incidence, results and effects of musculoskeletal pain in 9 regions of the body, including neck, shoulder, back, elbow, hand/wrist, waist, hip/thigh, knee, foot/ankle. . In this questionnaire, the age of onset of pain, hospitalization due to pain, changing the place of duty, having pain in the last year, last month and today are questioned. In addition, it is a questionnaire that can be filled by oneself or by interviewing the person, questioning whether the current pain affects the individual's work/home life, applying to a doctor/physiotherapist, taking medication and getting a report. Subjects are asked to mark the location of the pain on the body diagram. A high score indicates musculoskeletal pain.
Lower Extremity Functional Performance Evaluation Single Leg Jump Test | 5 months
  Individuals' lower extremity functional performance will be evaluated with the Single Leg Jump Test (TBS). TBST validity and reliability were reported as 0.85 with ICC ratio. For the test, 2 measuring tapes are affixed to the plastic rods at an angle of 180 degrees and it is requested to stand on the dominant foot with the tip of the toe to the starting point of the tape measure. While the individual is standing on the dominant right leg, the other leg is bent at the knee and asked to jump forward and the point where the individual falls (finger tip) is marked. Care should be taken to keep the hands on the waist while jumping. If he loses his balance while falling to the ground and gets support from the other foot, the test is considered invalid and repeated. Jumping was repeated 3 times for both extremities. Jump distance is calculated by measuring with a tape measure in centimeters and taking the average value.
Closed Kinetic Chain Upper Extremity Stability Test | 5 months
  The reliability of the Closed Kinetic Chain Upper Extremity Stability Test was determined by Oliveira et al. made by Dynamic stability of the shoulder will be evaluated with KKZÜEST. The tester first explains the test position to the athlete, then the test is started with the 'start' command and the test is finished with the 'stop' command. After the instructions and demonstration, 3 attempts are made to teach the test and 5 seconds rest between each attempt. Subjects will be placed in a push-up position with their hands 36 inches (91.44 centimeters) apart on 1.5 inches (3.81 centimeters) wide strips. While one hand is fixed on the ground, it is asked to raise the other hand, touch the band under the fixed hand and take it back to the starting point. The same movement is repeated for the opposite side and 15 seconds. The number of repetitions performed in the test is recorded. The average of 3 repetitions of the test is taken.
Closed Kinetic Chain Lower Extremity Stability Test | 5 months
  Closed Kinetic Chain Lower Extremity Stability Test, Arıkan et al. Its reliability and validity were made in 2021 by The test was developed to measure trunk and lower extremity strength, strength and stability of the whole body. In order to teach the test from the instructions and demonstration, 3 trials are made and 5 seconds rest between each trial. Starting position, the person is on his forearms with feet shoulder-width apart, toes in contact with the floor, and body lying in a straight line. While maintaining the starting position of the body, the individual is asked to bring one foot to the diagonal outer side of the other foot. After touching the side of the other foot, the foot returns to the starting position. Then the person performs the same movement with the other foot. The number of repetitions in 15 seconds is recorded as in the closed kinetic chain upper extremity stability test. The average of 3 repetitions of the test is taken.
Upper Extremity Y Balance Test | 5 months
  The Upper Extremity Y Balance Test is used to determine the risk of injury in musculoskeletal problems. Explains the test position to the athlete, then makes 3 attempts to teach the test and rests for 5 seconds between each attempt. The measurement is started with the subject both hands shoulder-width apart, right hand on the stance plate, and left hand on the access cursor. By maintaining the push-up position, the distance reached with the left hand is recorded in 3 directions, first medial, then inferolateral and finally superolateral. The person returns to the starting point in a controlled manner without changing his position. Tests are repeated 3 times on both extremities. Upper extremity length to be used in scoring is determined by measuring the distance between cervical C7 and the longest fingertip with a tape measure.
Lower Extremity Y Balance Test | 5 months
  The tester first explains the test position to the athlete, then three trials are made in order to teach the test, and after each trial, it is rested for 5 seconds. In the test setup, 3 measuring tapes are attached to the plastic bars at an angle of 135 degrees. Individuals stand on one leg at the intersection of the three measuring tapes. The fingertip is asked to extend in the anterior, posteromedial and posterolateral directions. Care is taken that the individual does not lose his balance by placing his hands on his waist, and that the heel of the foot he is standing on does not rise from the ground. The test is repeated 3 times in each direction. The length of the lower extremity (between the spina iliaca anterior superior and the medial 3malleolus) will be measured with a tape measure.
Posture Evaluation | 5 months
  Posture of the athletes in lateral and squat positions was reported by Hopkins et al. It will be measured with the PostureScreen Mobile® Application, of which validity and reliability study has been done by. Postures of the athletes in lateral and squat positions will be done on the smartphone using the PostureScreen Mobile® App. The specific points determined in the application for the lateral and squat positions of the athletes will be marked using the touch screen on the photographs taken, and according to these points, the postural disorder values and the degree of the disorder will be calculated and reported for each variable in cm or degrees via the software.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Paksoy, Bachelor, Principal Investigator — Eastern Mediterranean University; Berkiye Kırmızıgil, Associate Professor, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Mersin, Famagusta, Turkey (Türkiye)

REFERENCES:
- [Background] Claudino JG, Gabbett TJ, Bourgeois F, Souza HS, Miranda RC, Mezencio B, Soncin R, Cardoso Filho CA, Bottaro M, Hernandez AJ, Amadio AC, Serrao JC. CrossFit Overview: Systematic Review and Meta-analysis. Sports Med Open. 2018 Feb 26;4(1):11. doi: 10.1186/s40798-018-0124-5. PMID 29484512
- [Background] Angel Rodriguez M, Garcia-Calleja P, Terrados N, Crespo I, Del Valle M, Olmedillas H. Injury in CrossFit(R): A Systematic Review of Epidemiology and Risk Factors. Phys Sportsmed. 2022 Feb;50(1):3-10. doi: 10.1080/00913847.2020.1864675. Epub 2021 Jan 7. PMID 33322981
- [Background] Alaca N, Safran EE, Karamanlargil AI, Timucin E. Translation and cross-cultural adaptation of the extended version of the Nordic musculoskeletal questionnaire into Turkish. J Musculoskelet Neuronal Interact. 2019 Dec 1;19(4):472-481. PMID 31789298
- [Background] Forthomme B, Dvir Z, Crielaard JM, Croisier JL. Isokinetic assessment of the shoulder rotators: a study of optimal test position. Clin Physiol Funct Imaging. 2011 May;31(3):227-32. doi: 10.1111/j.1475-097X.2010.01005.x. Epub 2011 Jan 13. PMID 21470363
- [Background] Fifolato TM, Nardim HCB, do Carmo Lopes ER, Suzuki KAK, da Silva NC, de Souza Serenza F, Fonseca MCR. Association between muscle strength, upper extremity fatigue resistance, work ability and upper extremity dysfunction in a sample of workers at a tertiary hospital. BMC Musculoskelet Disord. 2021 Jun 1;22(1):508. doi: 10.1186/s12891-021-04256-y. PMID 34074292
- [Background] Arikan H, Maras G, Akaras E, Citaker S, Kafa N. Development, reliability and validity of the Closed Kinetic Chain Lower Extremity Stability Test (CKCLEST): a new clinical performance test. Res Sports Med. 2022 Sep-Oct;30(5):475-490. doi: 10.1080/15438627.2021.1906674. Epub 2021 Mar 24. PMID 33759654
- See also: 1 — http://dergipark.org.tr/en/download/article-file/925714
- See also: 17 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3325634/pdf/ijspt-07-139.pdf
- See also: 18 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2953327/pdf/najspt-04-092.pdf
- See also: 19 — http://scholarsarchive.byu.edu/cgi/viewcontent.cgi?article=5118&context=etd